CLINICAL TRIAL: NCT02834624
Title: Comparison of Curosurf and Infasurf in the Treatment of Preterm Infants With Respiratory Distress Syndrome
Acronym: NEOSURF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1206415
Record Dates: First submitted 2016-05-19; First posted 2016-07-15 (Estimated); Results first posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-05

CONDITIONS: Respiratory Distress Syndrome
Keywords: surfactant; respiratory distress syndrome; inflammation; c-reactive protein; lipid peroxidation
MeSH Terms: conditions — Respiratory Distress Syndrome; Inflammation | interventions — poractant alfa; calfactant

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Calfactant (Active Comparator): Randomized to receive Infasurf as the surfactant to treat respiratory distress syndrome. Doses 3ml/kg. to be repeated as needed by determination of attending neonatologist.
  Interventions: Drug: calfactant
- Poractant Alfa (Active Comparator): Randomized to receive Curosurf as the surfactant to treat respiratory distress syndrome. Doses 3ml/kg. to be repeated as needed by determination of attending neonatologist.
  Interventions: Drug: Poractant alfa

INTERVENTIONS:
Drug: Poractant alfa — Randomized to receive Curosurf as the surfactant to treat respiratory distress syndrome. Doses 3ml/kg. to be repeated as needed by determination of attending neonatologist.
  Other Names: Curosurf
  Arms: Poractant Alfa
Drug: calfactant — Randomized to receive Infasurf as the surfactant to treat respiratory distress syndrome. Doses 3ml/kg. to be repeated as needed by determination of attending neonatologist
  Other Names: Infasurf
  Arms: Calfactant

SUMMARY:
Premature infants frequently have trouble breathing after birth. If the respiratory disorder is caused by surfactant deficiency or dysfunction, the disease is treated with a medication called surfactant that is given to the infant through a tube inserted into the windpipe. This study will compare the safety of two of the commonly used surfactants, poractant and calfactant,in the United States. Poractant has added chemicals called phospholipids which are known to cause inflammation and irritation in the body of premature infants. The investigators will compare this to another similar surfactant that does not contain these chemicals by looking at samples from the windpipe, while the tube is in place, and from blood tests in the first few days of life.

The investigators are hoping to learn whether calfactant is a safer therapeutic agent to treat respiratory distress syndrome in preterm infants compared to poractant.

DETAILED DESCRIPTION:
30 infants were randomized to receive either poractant or calfactant for Respiratory Distress Syndrome.

Tracheal aspirates were obtained to look for increase in macrophage and blood samples were drawn to look for markers of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled prior to delivery with signed informed consent and HIPAA by parents
* Gestational age of less than 35 weeks
* No maternal chorioamnionitis of other maternal or fetal infection
* Respiratory Distress Syndrome (RDS) determined by the attending neonatologist that needs to be treated with exogenous surfactant and mechanical ventilation

Exclusion Criteria:

* Major Birth Defect, Malformation Syndrome
* Chromosomal or Inherited Metabolic Disorder
* Proven Presence of an Immunodeficiency
* Antenatal exposure of illicit substance (e.g., methamphetamines, cocaine, etc., but not marijuana)
* Birth Asphyxia (cord pH <7.0, Apgar score of 3 or less at 10 minutes of age)
* HIV or other congenital viral, bacterial or fungal infection
* Lack of Parental consent of refusal of attending neonatologist to allow participation
* Discretion of the investigator
* The legal representative of the infant or the patient's primary physician are not committed to providing full, aggressive life support

Ages: 22 Weeks to 35 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2013-07; Primary Completion 2015-02 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Naomi Lauriello, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri, Women's and Children's Hospital, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Infants < 35 weeks gestation requiring intubation and surfactant for Respiratory Distress Syndrome. Infants with suspected congenital infection, major birth defects, known chromosomal disorder, cord blood pH < 7.0, or Apgar score of 3 or < at 10 minutes were excluded. The infants were randomized to receive either Poractant or Calfactant.
Groups:
- Poractant: Randomized to receive poractant alfa (Curosurf) as the surfactant to treat respiratory distress syndrome. Doses 3ml/kg. to be repeated as needed by determination of attending neonatologist.
- Calfactant: Randomized to receive calfactant (Infasurf) as the surfactant to treat respiratory distress syndrome. Doses 3ml/kg. to be repeated as needed by determination of attending neonatologist.
Period: Overall Study
Arm/Group | Poractant | Calfactant
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Preterm infants less than 35 weeks gestation who required intubation for RDS and surfactant administration
Groups:
- Total: Total of all reporting groups
Arm/Group | Poractant | Calfactant | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 15 | 15 | 30
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Unknown | 15 | 15 | 30
Region of Enrollment [Number; unit: participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Blood C-reactive (CRP) Protein
Description: Difference between measurement of CRP at baseline and 48 hours after administration of surfactant
Time Frame: baseline, 48 hours
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Poractant | Calfactant
Number analyzed (Participants) | 15 | 15
mg/dL | 1.300 (1.644) | 0.193 (0.337)
Statistical Analysis 1: Comparison: Poractant vs Calfactant; Sample size calculations used a Chi-square for independence, u = 1, p =.05, power = .80, effect size = .60, which required 22 total subjects; Test type: Other; p < .05, t-test, 1 sided

2. Secondary Outcome: Presence of Pulmonary Hemorrhage
Description: Significant and Persistent Blood present in the trachea during endotracheal tube suctioning.
Time Frame: intraoperative
Population: This data is unavailable from the research department as it was not collected.
Arm/Group | Poractant | Calfactant
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Number of Tracheal Macrophages
Description: measurement of lipid peroxidation in tracheal aspirate samples and cytology of tracheal aspirates.in tracheal aspirate
Time Frame: baseline, 48 hours
Measure: Mean (Standard Deviation); unit: white cells/high-powered field
Arm/Group | Poractant | Calfactant
Number analyzed (Participants) | 15 | 15
white cells/high-powered field | 2.3 (1.8) | 2.0 (1.2)
Statistical Analysis 1: Comparison: Poractant vs Calfactant; Test type: Other; p = 0.63, t-test, 1 sided

ADVERSE EVENTS:
Arm/Group | Calfactant | Poractant Alfa
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes